CLINICAL TRIAL: NCT05403307
Title: A Real-world Evidence Study of BNT162b2 mRNA Covid-19 Vaccine Among Children Aged 5 to 11 Years in Brazil
Brief Title: A Real-world Evidence Study of BNT162b2 mRNA Covid-19 Vaccine Among Children in Brazil
Status: Completed | Type: Observational
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Universidade Federal do Paraná (Other); Pfizer (Industry); Inova Medical (Other)
Responsible Party: Sponsor
Other Study IDs: BNT162b2 pediatric Toledo
Record Dates: First submitted 2022-05-27; First posted 2022-06-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (7):
- Two doses or more of BNT162b2: Defined as ≥ 2 doses of BNT162b2 COVID-19 vaccine received with ≥7 days between receipt of the 2nd dose and acute respiratory illness (ARI) symptom onset. This group will serve as the 'exposed' group evaluated in the primary objective.
  Interventions: Biological: Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine
- One dose of BNT162b2: Defined as 1 dose (only) of Pfizer/BioNTech BNT162b2 COVID-19 vaccine received with ≥14 days between receipt of the 1st dose and ARI symptom onset.
  Interventions: Biological: Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine
- One dose or more of BNT162b2: Defined as ≥1 dose of Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine received with ≥14 days between receipt of the 1st dose and ARI symptom onset.
  Interventions: Biological: Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine
- Two doses of BNT162b2: Defined as 2 doses of BNT162b2 COVID-19 vaccine received with ≥7 days between receipt of the 2nd dose and acute respiratory illness (ARI) symptom onset.
  Interventions: Biological: Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine
- Three doses of BNT162b2: Defined as 3 doses of BNT162b2 COVID-19 vaccine received with ≥7 days between receipt of the 3rd dose and acute respiratory illness (ARI) symptom onset.
  Interventions: Biological: Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine
- Fully vaccinated with other available COVID-19 vaccines: Defined as fully vaccinated with available COVID-19 vaccines according to Brazil National Immunization Program recommendations.
  Interventions: Biological: CoronaVac COVID-19 vaccine
- Never vaccinated: Defined as never received any COVID-19 vaccine. This group will serve as the reference exposure group (i.e., 'unexposed' group) in all vaccine effectiveness analyses.

INTERVENTIONS:
Biological: Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine — Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine
  Groups: One dose of BNT162b2; One dose or more of BNT162b2; Three doses of BNT162b2; Two doses of BNT162b2; Two doses or more of BNT162b2
Biological: CoronaVac COVID-19 vaccine — CoronaVac COVID-19 vaccine
  Groups: Fully vaccinated with other available COVID-19 vaccines

SUMMARY:
The present test-negative design study aims to estimate the real-world effectiveness of Pfizer-BioNTech BNT162b2 mRNA vaccine on symptomatic SARS-CoV-2 infection and its consequences among children aged 5 to 11 years in the city of Toledo in Southern Brazil.

Individuals aged 5 to 11 years who seek the public healthcare system with symptoms suggestive COVID-19 will be enrolled. Participants with a positive reverse transcriptase polymerase chain reaction (RT-PCR) test for SARS-CoV-2 will be classified as cases, and those with negative RT-PCR test for SARS-CoV-2 will be classified as controls. Cases will be followed-up for a period of 3 months by means of structured telephone interviews.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 11 years;
* Resident of Toledo city;
* Seeking care in the public healthcare system with symptoms suggestive of COVID-19 defined as follows: 1) ARI symptoms (nasal congestion, rhinorrhea, anosmia, sore throat, hoarseness, new or increased-from-baseline cough, sputum production, dyspnea, wheezing, myalgia) OR 2) Admitting diagnosis suggestive of ARI (pneumonia, upper respiratory infection, bronchitis, influenza, cough, asthma, viral respiratory illness, respiratory distress, AND/OR respiratory failure).
* Nasal or nasopharyngeal sample for SARS-CoV-2 test obtained as standard of care.

Exclusion Criteria:

* SARS-CoV-2-directed antiviral treatment within the past 30 days;
* COVID-19 monoclonal antibody therapy within the past 90 days;
* COVID-19 convalescent serum therapy within the past 90 days;
* Failure to perform RT-PCR for diagnosis of SARS-CoV-2 infection.

Ages: 5 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: The present study population will be composed by individuals aged 5 to 11 years who seek the public healthcare system of Toledo city with symptoms suggestive COVID-19. Participants with a positive RT-PCR test for SARS-CoV-2 will be classified as cases, and those with negative RT-PCR test for SARS-CoV-2 will be classified as controls.
Sampling Method: Non-Probability Sample
Enrollment: 757 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Odds of symptomatic SARS-CoV-2 infection | At the moment of enrollment
  Odds of symptomatic SARS-CoV-2 infection defined by the presence of symptoms suggestive COVID-19 with a positive RT-PCR test for SARS-CoV-2. Symptoms suggestive of COVID-19 are defined as follows: 1) Acute respiratory illness symptoms (nasal congestion, rhinorrhea, anosmia, sore throat, hoarseness, new or increased-from-baseline cough, sputum production, dyspnea, wheezing, myalgia) OR 2) Admitting diagnosis suggestive of ARI (pneumonia, upper respiratory infection, bronchitis, influenza, cough, asthma, viral respiratory illness, respiratory distress, AND/OR respiratory failure).

SECONDARY OUTCOMES:
Odds of symptomatic SARS-CoV-2 infection due to Omicron variant | At the moment of enrollment
  Odds of symptomatic SARS-CoV-2 infection due to Omicron variant defined by the presence of symptoms suggestive COVID-19 with a positive RT-PCR test for SARS-CoV-2 Omicron variant
Odds of symptomatic SARS-CoV-2 infection due to other circulating variants of concern | At the moment of enrollment
  Odds of symptomatic SARS-CoV-2 infection due to other circulating variants of concern defined by the presence of symptoms suggestive COVID-19 with a positive RT-PCR test for SARS-CoV-2 variants of concern.
Duration of COVID-19 symptoms | within 90 days from enrollment
  Length of COVID-19-related symptoms
Incidence of hospitalization due to COVID-19 | Within 90 days from enrollment
  Incidence of hospital admission due to COVID-19
Incidence of PICU admission | Within 90 days from enrollment
  Incidence of Pediatric intensive care unit admission
Incidence of invasive mechanical ventilation | Within 90 days from enrollment
  Incidence of invasive mechanical ventilation
Incidence of multisystem inflammatory syndrome | Within 90 days from enrollment
  Incidence of multisystem inflammatory syndrome
Mortality due to COVID-19 | Within 90 days from enrollment
  Incidence of COVID-19-related mortality
Prevalence of long COVID-19 symptoms at 3 months | Within 90 days from enrollment
  Prevalence of long COVID-19-related symptoms (fatigue, muscular weakness, dyspnea, cough, loss of taste or smell, concentration or memory difficulties, sleep disorders, headache)

CONTACTS AND LOCATIONS:
Overall Officials: Regis G Rosa, MD, PhD, Principal Investigator — Hospital Moinhos de Vento, INOVA; Maicon Falavigna, MD, PhD, Principal Investigator — Hospital Moinhos de Vento, INOVA
Locations (5):
- Brazil (5):
  - Jardim Coopagro, Toledo, Paraná
  - Jardim Cosmos primary healthcare unit, Toledo, Paraná
  - Jardim Maracanã, Toledo, Paraná
  - Jardim Porto Alegre, Toledo, Paraná
  - Pediatric Emergency Service, Toledo, Paraná

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodrigues CO, Spinardi J, Rosa RG, Falavigna M, de Souza EM, Manfio JL, de Souza AP, de Araujo CLP, Cohen M, Barbosa GRGDV, Silva FKR, Sganzerla D, da Silva MMD, Ferreira D, Kunkel NT, Camargo NI, Sarturi JC, Guilhem MC, de Oliveira JC, Lopes CC, Widmar F, Barufi LK, da Silva GN, Gradia DF, Brandalize APC, Royer CA, Luiz RM, Baura VA, Abreu H, Poitevin CG, Kucharski GA, Pedrotti F, Valluri SR, Srivastava A, Juliao VW, Melone OC, Allen KE, Kyaw MH, Castillo GDCM, McLaughlin JM; Toledo BNT162b2 Study Group Investigators. Real-world effectiveness of original BNT162b2 mRNA COVID-19 against symptomatic Omicron infection among children 5-11 years of age in Brazil: A prospective test-negative design study. Immunol Lett. 2024 Oct;269:106903. doi: 10.1016/j.imlet.2024.106903. Epub 2024 Jul 26. PMID 39069096